CLINICAL TRIAL: NCT04440085
Title: RANDOMIZED CASE-CONTROLLED TRIAL ASSESSING MIDODRINE (GUTRON®) IN POSTOPERATIVE VASOPLEGIC PATIENTS
Brief Title: RaGuS Trial by Postoperative Patients
Acronym: RaGuS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bürgerspital Solothurn (Other)
Responsible Party: Principal Investigator, Marcos Delgado, Principal investigator, Bürgerspital Solothurn
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: RaGuS
Record Dates: First submitted 2020-06-13; First posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Vasoplegic Syndrome; Sirs Due to Noninfectious Process Without Organ Dysfunction; Orthostatic Hypotension
Keywords: Midodrine; Vasoplegic syndrome; Noradrenaline; SIRS
MeSH Terms: conditions — Vasoplegia; Hypotension, Orthostatic | interventions — Midodrine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, single-center, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Midodrine will be administered every 8 hours, increasing the dose gradually until a maximum of 30 mg a day is reached. It will be given orally in the following sequence: 2.5 mg - 5 mg - 7.5 mg - 10 mg. The target standard perfusion pressure for all the patients will be a mean arterial pressure (MAP) > 65 mmHg, with unchanged dose of midodrine after target pressure is reached. If the pressure continues to increase, the same sequence will be followed for dose de-escalation.
  Interventions: Drug: Midodrine Hydrochloride
- Control group (Placebo Comparator): By placebo group will be followed the same strategy.The target standard perfusion pressure for all the patients will be a mean arterial pressure (MAP) > 65 mmHg, with unchanged dose of placebo after target pressure is reached. If the pressure continues to increase, the same sequence will be followed for dose de-escalation.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Midodrine Hydrochloride — All patients become standard care resuscitation treatment using liquids and vasoactive drugs in order to get a median arterial pressure ≥ 65 mmHg. Midodrine will be administered according to the evolution of the patient's mean pressure.
  Arms: Intervention group
Drug: Placebo — All patients become standard care resuscitation treatment using liquids and vasoactive drugs in order to get a median arterial pressure ≥ 65 mmHg. Placebo will be administered according to the evolution of the patient's mean pressure.
  Arms: Control group

SUMMARY:
Vasoplegic syndrome is characterized clinically by reduced systemic vascular resistance and normal or increased cardiac output. It is principally observed in cardiovascular and orthopedic interventions and is characterized by a systemic inflammatory response with the inability of the vascular endothelial muscles to contract and a resistance to the action of vasoactive drugs. This event extends the length of stay in the critical care area due to the need of vasoactive drugs.

The investigators aim to assess the standardized application of midodrine in postoperative patients without sepsis and need of vasoactive drugs in order to reduce the length of stay in critical care area and for extension in hospital.

DETAILED DESCRIPTION:
Midodrine is an alpha 1 receptor agonist used usually in cases of hypotension helping to increase blood pressure. The main indication is orthostatic hypotension but there are other clinical conditions where this medicament is often used like hypotension by dialysis, hepatorenal syndrome and after carotid artery stenting.

Vasoplegic syndrome coul be interpreted as a variant of orthostatic hypotension that happens usually after surgical interventions. It produces a loss of systemic vascular resistance due to inflammatory reaction without any signs of infection.

The investigators aim to conduct a randomized, double-blind, single-center, placebo-controlled study of midodrine in patients who present postoperative vasoplegia with no active signs of sepsis but need of vasoactive drugs (Noradrenalin).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Need of vasoactive drugs after three hours from arrival and adequate volume recovery.

Exclusion Criteria:

* Signs of infection (anamnesis or pro-calcitonin > 0.2 with leukocytosis, CRP and/or fever)
* Serum lactate > 2mmol/l
* Mechanical ventilation
* Therapeutic restrictions or comfort measures at arrival
* "de novo" or acute on chronic heart failure (Reduction of known ejection fraction for more than 20 percent, signs of acute lung edema)
* Pregnant
* Patients with digoxin treatment or history of glaucoma.
* History of midodrine allergy, pheochromocytoma, thyrotoxicosis, tachyarrhythmias or ventricular fibrillation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-14 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-14 (Estimated)

PRIMARY OUTCOMES:
Time | aproximately 2 days
  Hours from initiation of treatment with midodrine to discharge from critical care area

SECONDARY OUTCOMES:
Length of stay | aproximately 7 days
  days in critical care area and hospital
Vasopresors | aproximately 2 days
  Noradrenalin needed doses
Fluid balance | aproximately 2 days
  cumulative fluid balance in mililiter

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Delgado, MD, Principal Investigator — Bürgerspital Solothurn

IPD SHARING:
Plan to Share IPD: No
We have decided for the Trial not to share the participant Information.

REFERENCES:
- [Result] Tchen S, Sullivan JB. Clinical utility of midodrine and methylene blue as catecholamine-sparing agents in intensive care unit patients with shock. J Crit Care. 2020 Jun;57:148-156. doi: 10.1016/j.jcrc.2020.02.011. Epub 2020 Feb 19. PMID 32145658
- [Result] Shaefi S, Mittel A, Klick J, Evans A, Ivascu NS, Gutsche J, Augoustides JGT. Vasoplegia After Cardiovascular Procedures-Pathophysiology and Targeted Therapy. J Cardiothorac Vasc Anesth. 2018 Apr;32(2):1013-1022. doi: 10.1053/j.jvca.2017.10.032. Epub 2017 Oct 27. PMID 29223724
- [Result] Jans O, Mehlsen J, Kjaersgaard-Andersen P, Husted H, Solgaard S, Josiassen J, Lunn TH, Kehlet H. Oral Midodrine Hydrochloride for Prevention of Orthostatic Hypotension during Early Mobilization after Hip Arthroplasty: A Randomized, Double-blind, Placebo-controlled Trial. Anesthesiology. 2015 Dec;123(6):1292-300. doi: 10.1097/ALN.0000000000000890. PMID 26492477
- [Result] Smits M, Lin S, Rahme J, Bailey M, Bellomo R, Hardidge A. Blood Pressure and Early Mobilization After Total Hip and Knee Replacements: A Pilot Study on the Impact of Midodrine Hydrochloride. JB JS Open Access. 2019 May 14;4(2):e0048. doi: 10.2106/JBJS.OA.18.00048. eCollection 2019 Apr-Jun. PMID 31334462
- [Result] Levine AR, Meyer MJ, Bittner EA, Berg S, Kalman R, Stanislaus AB, Ryan C, Ball SA, Eikermann M. Oral midodrine treatment accelerates the liberation of intensive care unit patients from intravenous vasopressor infusions. J Crit Care. 2013 Oct;28(5):756-62. doi: 10.1016/j.jcrc.2013.05.021. Epub 2013 Jul 8. PMID 23845791
- [Result] Cardenas-Garcia JL, Whitson MR, Healy K, Koenig S, Narasimhan M, Mayo P: Safety of oral midrodrine as a mehtod of weaning from intravenous vasoactive medication in the medical intensive care unit. Chest 2014, 146(4):224A.
- [Result] Rizvi MS, Nei AM, Gajic O, Mara KC, Barreto EF. Continuation of Newly Initiated Midodrine Therapy After Intensive Care and Hospital Discharge: A Single-Center Retrospective Study. Crit Care Med. 2019 Aug;47(8):e648-e653. doi: 10.1097/CCM.0000000000003814. PMID 31107279
- [Result] Whitson MR, Mo E, Nabi T, Healy L, Koenig S, Narasimhan M, Mayo PH. Feasibility, Utility, and Safety of Midodrine During Recovery Phase From Septic Shock. Chest. 2016 Jun;149(6):1380-3. doi: 10.1016/j.chest.2016.02.657. Epub 2016 Mar 4. PMID 26953217
- [Result] Anstey MH, Wibrow B, Thevathasan T, Roberts B, Chhangani K, Ng PY, Levine A, DiBiasio A, Sarge T, Eikermann M. Midodrine as adjunctive support for treatment of refractory hypotension in the intensive care unit: a multicenter, randomized, placebo controlled trial (the MIDAS trial). BMC Anesthesiol. 2017 Mar 21;17(1):47. doi: 10.1186/s12871-017-0339-x. PMID 28327122